CLINICAL TRIAL: NCT07052955
Title: The Effect of Health Riddles on Fear, Anxiety, and Pain in Circumcised Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gümüşhane Universıty (Other)
Responsible Party: Principal Investigator, Hatice Oğuzhan, Lecturer, Gümüşhane Universıty
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Health Riddles in Pediatry
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Circumcision, Male
Keywords: Child; anxiety; fear; pain; circumcision; health riddles
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive routine clinical care. No intervention will be made.
- Experimental Group (Experimental): Before the circumcision, children will be shown a video animation show and will be made to play games with health riddles and normal riddle books.
  Interventions: Other: The Normal Riddles Book; Other: Health Riddles Group

INTERVENTIONS:
Other: The Normal Riddles Book — The distribution of the participating children to the experimental and control groups will be carried out by simple random sampling method. Children included in the Normal Riddle Book group will be introduced to a book containing general, entertaining riddles that are not related to health during the pre-circumcision period.
  The book will be given to the children approximately 1 hour before the circumcision operation and the children will be allowed to read the puzzles, solve them or interact with the researcher/nurse. The application period is planned as approximately 20-30 minutes.
  The children's fear, anxiety and pain levels will be measured before and after the application. During the application process, the children's attention level, interest in the book and general behavior will be observed and recorded.
  Arms: Experimental Group
Other: Health Riddles Group — The children included in this group will be presented with the Health Riddles Book, which contains health information and is prepared to reduce fear and anxiety before the circumcision.
  The book will be given to the children approximately 1 hour before the circumcision procedure and the children will be allowed to read the riddles or interact with the researcher/nurse. The application time is planned to be 20-30 minutes. Before and after the application, the children's fear, anxiety and pain levels will be measured with the Introductory Information Form, Child Fear Scale, Child Anxiety Scale-State and Wong-Baker Face Pain Scale.
  The data obtained from the health riddles group will be compared with the data obtained from the normal riddle and control groups and the unique effect of the riddles containing health information on fear, anxiety and pain will be analyzed.
  Arms: Experimental Group

SUMMARY:
This study was designed as a randomized controlled experimental method to examine the effects of health puzzles on the fear, anxiety and pain levels that occur in the pre- and postoperative periods in children who underwent circumcision.

DETAILED DESCRIPTION:
In the study, children aged 4-6 who came to be circumcised were divided into three groups: the Normal Circumcision Control Group, which received standard care and information, the Normal Riddle Group, which was supported by general fun riddles that did not contain health content, and the Health Riddles Group, which received an intervention that included health information and aimed to reduce children's fear and anxiety levels. The children's fear, anxiety and pain levels before and after the surgery will be measured using the Introductory Information Form, the Children's Fear Scale, the Children's Anxiety Scale-State and the Wong-Baker Facial Pain Scale as data collection tools.

ELIGIBILITY:
Inclusion Criteria:

* Children who apply to Gümüşhane State Hospital Pediatric Surgery Department for circumcision
* Children between the ages of 4-6
* Not having had any previous surgical intervention
* Not having any problems with vision, hearing or speech
* Written consent given by a parent or legal guardian
* Not having health problems that could affect the research results, such as chronic disease or developmental delay
* The child and his/her family being open to communication and willing to cooperate during the study participation process

Exclusion Criteria:

* If the child or family does not want to continue the research
* If there is a sudden and serious deterioration in the child's health
* If participants do not comply with the research protocol, do not use the provided materials or do not participate in the measurements and do not continue
* If unexpected complications develop during the circumcision procedure
* If it is determined that the rights of the participants have been violated in accordance with ethical rules
* In these cases, the participant will be removed from the research and appropriate health care will be provided where necessary.

Ages: 4 Years to 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male
Enrollment: 120 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-11-10 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | Baseline
  The introductory information form prepared by the researchers consists of items related to the child's age, gender, height, weight, place of residence, number of siblings, previous hospitalization, previous surgery, mother's age, education status, father's age, education status and the family's economic status.
Child Fear Scale (CFS) | Baseline and up to 4 weeks
  This scale was developed by McMurtry and colleagues in 2011 and was adapted to Turkish by Gerçeker and his team in 2018 and validated. Designed for children between the ages of 5 and 10, this scale presents facial muscle changes in fearful expressions with a graphic artist's drawings based on photographs of frightened faces. The scale can be used by the family, child, or researcher to evaluate children. The scale shows the child a scale containing five facial expressions scored between 0 and 4. These expressions are interpreted as follows: 0: Neutral expression (no fear), 1: Very little fear, 2: Some fear, 3: More fear, 4: Highest level of fear. This scale can be used to measure the child's level of fear before and during the procedure.
Child Anxiety Scale-State (CAS-D) | Baseline and up to 4 weeks
  The "Child Anxiety Scale-State" (CAS-D) scale, developed by Ersig and his colleagues in 2013, is used to measure the situational anxiety of children between the ages of 4-10. Its validity was provided by Gerçeker and his team in 2018. CAS-D is designed in the shape of a thermometer and has a bulb chamber at the bottom and horizontal lines upwards. Each horizontal line represents one point, and there are 10 points in total. The bottom line represents a score of 0 and indicates a situation where there is no anxiety. The anxiety level increases as you go higher, and the top line represents the highest anxiety with a score of 10.
Wong Baker Pain Rating Scale | Baseline and up to 4 weeks
  The Wong-Baker Faces Pain Rating Scale is an adaptation of the Faces Rating Scale, a picture projection technique that uses 6 pictures of a child's facial expressions in pain to assess the child's level of pain. This scale is used to best describe the child's current level of pain.
  The child is asked to choose the face that best describes their pain. The descriptions of the faces are as follows:
  Face 0: Depicts a painless, happy face, meaning "I'm very happy, I'm in no pain." Face 5: Depicts a crying face, meaning "it hurts as much as you can imagine, but you don't have to cry to feel that bad." The responses on this 5-point scale range from 0 (very happy, no pain) to 5 (it hurts as much as you can imagine) and help determine the child's level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice OĞUZHAN, 1, Principal Investigator — Gümüşhane Universıty
Locations (1):
- Baglarbasi District Shahbenders District Cluster Houses No.56/B Center/Gumushane, Gümüşhane, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuncay S, Tufekci FG. The effect of nursing interventions with therapeutic play and video animations prepared with psychodrama technique in reducing fear, anxiety, and pain of children at male circumcision: A randomized controlled study. Int J Urol. 2023 Jul;30(7):592-599. doi: 10.1111/iju.15184. Epub 2023 Mar 31. PMID 36999456
- See also: Randomized Controlled Trial — https://pubmed.ncbi.nlm.nih.gov/36999456/